CLINICAL TRIAL: NCT02339064
Title: A Phase 3, Open-Label Study of the Safety, Efficacy and Tolerability of Apomorphine Administered by Continuous Subcutaneous Infusion in Advanced Parkinson's Disease Patients With Unsatisfactory Control on Available Therapy
Brief Title: Infusion of Apomorphine: Long-term Safety Study
Acronym: INFUS-ON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MDD US Operations, LLC a subsidiary of Supernus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Supernus Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USWM-AP2-3000
Record Dates: First submitted 2014-03-31; First posted 2015-01-15 (Estimated); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease,; apomorphine; Apokyn; dopamine agonist; levodopa; advanced; PD; carbidopa; pramipexole; ropinirole; rotigotine; MAO-B inhibitors; COMT inhibitors; off; dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apomorphine infusion (Experimental): Continuous subcutaneous apomorphine infusion
  Interventions: Drug: apomorphine infusion

INTERVENTIONS:
Drug: apomorphine infusion — Treatment with apomorphine provided by continuous subcutaneous infusion using a portable external electronic pump device

SUMMARY:
This is a Phase 3, multicenter, open-label, safety and tolerability study of continuous apomorphine infusion in subjects with advanced Parkinson's Disease (PD) whose motor fluctuations remain unsatisfactory with levodopa (or levodopa/carbidopa) and at least one other class of drugs or mode of therapy for PD.

DETAILED DESCRIPTION:
This Phase 3, multicenter, open-label study will assess the long-term safety and tolerability of continuous subcutaneous infusion of apomorphine in advanced Parkinson's disease (PD) patients whose motor fluctuations remain unsatisfactory with levodopa (or levodopa/carbidopa) and at least one other class of drugs or mode of therapy for PD.

Further, this study will assess the clinical effectiveness of continuous apomorphine subcutaneous infusion in reducing "off" time in advanced PD patients and to assess the clinical effectiveness of continuous subcutaneous infusion of apomorphine in improving "on" time without resulting in an increase in troublesome dyskinesias.

ELIGIBILITY:
Inclusion Criteria:

* Advanced idiopathic PD consistent with UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria
* Overall motor control is unsatisfactory in the opinion of the Investigator and subject despite optimized treatment with available therapies, which must include a stable regimen of daily maintenance levodopa (or levodopa/carbidopa), and at least one of the following other classes of therapies:
* Dopamine agonists (note: APOKYN intermittent injection is not to be considered here)
* Monoamine oxidase B [MAO B] inhibitors
* Catechol-O-methyltransferase (COMT) inhibitors
* Deep brain stimulation (DBS)
* Levodopa/carbidopa intestinal gel surgery (Duopa, Duodopa)
* Other - amantadine at doses of up to 400 mg per day)
* Experiences "off" periods averaging ≥3.0 hours per waking day
* Other criteria will be discussed in detail with potential subjects by site Investigator

Exclusion Criteria:

* Planned surgical intervention for the treatment of Parkinson's disease during participation in the study
* History of hypersensitivity to apomorphine hydrochloride or any of the ingredients of APOKYN PFS, including sodium metabisulfite
* Known, suspected, or planned pregnancy or lactation.
* Recent history (within the previous 12 months) of alcohol or substance abuse
* History of impulsive/compulsive behaviors primarily associated with the use of dopamine agonists
* History of previously treated or current diagnosis of malignant melanoma
* Exhibits certain signs and symptoms of cardiovascular disease
* Other criteria will be discussed in detail with potential subjects by site Investigator

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent of daily "off" time during the waking day | Baseline Visit to Week 12

SECONDARY OUTCOMES:
Percent daily "on" time without troublesome dyskinesias during waking day | Baseline Visit to Week 12
Percent of daily "off" time during the waking day | Baseline Visit to Treatment Weeks 2, 4, 8, 20, 28, 36, 44, and 52; and all Treatment Extension Period Visits
Percent of daily "on" time without troublesome dyskinesias during the waking day | Baseline Visit to Treatment Weeks 2, 4, 8, 20, 28, 36, 44, and 52; and all Treatment Extension Period Visits
Percent of daily "on" time without dyskinesias | Baseline Visit to Treatment Weeks 2, 4, 8, 20, 28, 36, 44, and 52; and all Treatment Extension Period Visits
Unified Parkinson's Disease Rating Scale - Motor Score | Baseline Visit to Week 12
Clinical Global Impression of Severity (CGI-S) and Change (CGI-C) Scale | Baseline Visit to Treatment Weeks 2, 4, 8, 20, 28, 36, 44, and 52; and all Treatment Extension Period Visits
Patient Global Impression of Severity (PGI-S) and Change (PGI-C) Scale | Baseline Visit to Treatment Weeks 2, 4, 8, 20, 28, 36, 44, and 52; and all Treatment Extension Period Visits
Parkinson's Disease Questionnaire | Baseline Visit to Treatment Weeks 2, 4, 8, 20, 28, 36, 44, and 52; and all Treatment Extension Period Visits
United Parkinson's Disease Rating Scale - Activities of Daily Living Score | Baseline Visit to Treatment Weeks 2, 4, 8, 20, 28, 36, 44, and 52; and all Treatment Extension Period Visits
Proportion of responders | Baseline Visit to Treatment Weeks 2, 4, 8, 20, 28, 36, 44, and 52; and all Treatment Extension Period Visits
Frequency and total dose of average daily intermittent injection APOKYN for subjects on APOKYN treatment at study entry | Baseline Visit to Treatment Weeks 2, 4, 8, 20, 28, 36, 44, and 52; and all Treatment Extension Period Visits

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiera Ceresoli-Borroni, PhD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (16):
- United States (16):
  - Phoenix, Arizona
  - Loma Linda, California
  - Los Angeles, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Boca Raton, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - West Bloomfield, Michigan
  - Albany, New York
  - Cincinnati, Ohio
  - Portland VA Medical Center, Portland, Oregon
  - Philadelphia, Pennsylvania
  - Kirkland, Washington